CLINICAL TRIAL: NCT02323438
Title: A Randomized, Controlled Study to Assess Biomarkers of Tobacco Exposure and Nicotine Pharmacokinetics in Smokers After a 5-Day In-Clinic Confinement Switch to an Electronic Cigarette or Nicotine Gum
Brief Title: Assess Biomarkers of Tobacco Exposure and Nicotine Pharmacokinetics in Smokers After a 5-Day In-Clinic Confinement Switch to an Electronic Cigarette or Nicotine Gum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: R.J. Reynolds Vapor Company (Industry)
Collaborators: Davita Clinical Research (Industry); RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CSD1304
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Smoking
Keywords: biomarkers of tobacco exposure; exposure; tobacco; nicotine; nicotine gum; electronic cigarette; e-cig
MeSH Terms: conditions — Smoking; Vaping | interventions — Nicotine; Menthol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Usual Brand (UB) Cigarettes (Active Comparator): Usual Brand Cigarette
  Interventions: Other: Usual Brand Cigarette
- Electronic Cigarette #1 (Experimental): VUSE® (original flavor, 29 mg nicotine)
  Interventions: Other: Electronic Cigarette #1
- Electronic Cigarette #2 (Experimental): VUSE® (menthol flavor, 26 mg nicotine)
  Interventions: Other: Electronic Cigarette #2
- Leading U.S. Nicotine Gum (Experimental): 4 mg nicotine polacrilex gum
  Interventions: Other: Leading U.S. Nicotine Gum

INTERVENTIONS:
Other: Usual Brand Cigarette — Combustible cigarette brand style smoked most frequently by subject
  Other Names: UB Cigarette
  Arms: Usual Brand (UB) Cigarettes
Other: Electronic Cigarette #1 — Electronic cigarette
  Other Names: VUSE® Digital Vapor Cigarette (original flavor, 29 mg nicotine)
  Arms: Electronic Cigarette #1
Other: Electronic Cigarette #2 — Electronic cigarette
  Other Names: VUSE® Digital Vapor Cigarette (menthol flavor, 26 mg nicotine)
  Arms: Electronic Cigarette #2
Other: Leading U.S. Nicotine Gum — 4 mg nicotine polacrilex gum
  Arms: Leading U.S. Nicotine Gum

SUMMARY:
A single-center, randomized, controlled, switching, open-label, parallel cohort study. Smoking subjects will be confined to a clinic for 9 days. During their stay, baseline assessments during ad libitum smoking will occur for the first 3 days. Following baseline, subjects will be switched to either an Electronic Cigarette or Nicotine Gum, and post-product switch assessments will occur for 6 days.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an Informed Consent Form (ICF) and complete questionnaires written in English;
2. Generally healthy males or females, 21 to 60 years of age (inclusive);
3. Screening expired-air carbon monoxide (ECO) level ≥ 15 parts per million (ppm; sample taken 30 to 60 minutes after smoking a single UB cigarette);
4. Currently smokes combustible, filtered, nonmenthol or menthol cigarettes, 83 mm to 100 mm length;
5. Self-reports that cigarettes are the only tobacco or nicotine-containing product used within 30 days of the Screening Visit;
6. Self-reports at the Screening Visit smoking at least 10 cigarettes per day and inhaling the smoke for at least 6 months prior to the Screening Visit;
7. Response to Fagerström Test for Nicotine Dependence (FTND) Question 1 ("How soon after you wake up do you smoke your first cigarette?") is either "Within 5 minutes" or "6-30 minutes" at the Screening Visit;
8. Positive urine cotinine test at Screening and Enrollment;
9. Willing to switch from current cigarette to VUSE Digital Vapor Cigarettes or nicotine gum for 6 days during in-clinic confinement (nonmenthol smokers willing to switch to VUSE Original Digital Vapor Cigarettes or nicotine gum; menthol smokers willing to switch to VUSE Menthol Digital Vapor Cigarettes or nicotine gum);
10. Willing to abstain from tobacco and nicotine use for at least 12 hours twice during confinement;
11. Willing to not participate for 60 days poststudy in donation of blood samples or in any study that requires collection of blood samples;
12. Females of childbearing potential must be willing to use a form of contraception acceptable to the Investigator from the time of signing the ICF until Study Discharge or be surgically sterile for at least 90 days prior to the Screening Visit;
13. Able to safely perform the required study procedures, as determined by the Investigator.

Exclusion Criteria:

1. Clinically significant or unstable/uncontrolled acute or chronic medical conditions at screening, as determined by the Investigator, that would preclude a subject from participating safely in the study (eg, hypertension, asthma, or other lung disease, cardiac disease, neurological disease, or psychiatric disorders) based on screening assessments such as safety labs, medical history, and physical/oral examinations;
2. Self-reports or safety labs indicate diabetes;
3. Self-reports stomach ulcers;
4. At risk for heart disease, as determined by the Investigator;
5. Use of medicine for treatment of depression or asthma;
6. Systolic blood pressure of ≥ 150 mmHg or a diastolic blood pressure of ≥ 95 mmHg, measured after being seated for 5 minutes;
7. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (anti-HCV);
8. Hemoglobin level is < 12 g/dL at Screening:
9. History or presence of hemophilia or any other bleeding disorders:
10. History or presence of clotting disorders with concomitant use of anticoagulants (eg, clopidogrel [Plavix®], warfarin [Coumadin®, Jantoven®], and aspirin [> 325 mg/day]);
11. Given a whole blood donation within 8 weeks (≤ 56 days) prior to Enrollment;
12. Plasma donation within (≤) 7 days prior to Enrollment;
13. Weight of ≤ 110 pounds;
14. Poor peripheral venous access;
15. Postponing a decision to quit smoking (defined as planning a quit attempt within 30 days of Screening) to participate in this study;
16. Employed by a tobacco company, the clinical site, or handles unprocessed tobacco as part of his/her job;
17. Use of marijuana-based materials within 30 days prior to screening;
18. Use of any medication or supplement that aids smoking cessation, including but not limited to any NRT (eg, nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within 30 days of the Screening Visit;
19. Use of injectable forms of medication(s), with the exception of injectable forms of birth control that are not required to be administered during the study period.
20. Self-reports drinking more than 14 servings of alcoholic beverages per week (1 serving = 12 oz of beer, 6 oz of wine, or 1 oz of liquor);
21. Females who have a positive pregnancy test, are pregnant, breastfeeding, or intend to become pregnant during the course of the study;
22. Females ≥ 35 years of age currently using systemic, estrogen-containing contraception, or hormone replacement therapy;
23. A positive urine drug screen without disclosure of corresponding prescribed concomitant medication(s) at the Screening Visit or Enrollment;
24. A positive alcohol breathalyzer test at Screening or Enrollment;
25. Regularly exposed to solvent fumes or gasoline (eg, painter, gas station mini-mart employee, etc.);
26. Determined by the Investigator to be inappropriate for this study, including a subject who is unable to communicate or unwilling to cooperate with the clinical staff;
27. Unable or unwilling to participate in the in-clinic confinement for the full study duration (total of 9 days).

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Changes in biomarkers of tobacco exposure after a 5-day, in-clinic switch from usual brand (UB) cigarettes to an Electronic Cigarette or Nicotine Gum | 6 days
  Determine percent change in carboxyhemoglobin (COHb), after 5 days of randomized IP use compared to UB smoking
Nicotine pharmacokinetics with respect to initiation of in-clinic investigational product (IP) use following a 12-hour tobacco and nicotine abstinence | -5, -0.5, 3, 5, 7.5, 10, 15, 20, 30, 45, 60, 75, 90, 120, 150, 180, 240, 300, 360 minutes
  Determine area under the plasma nicotine concentration versus time curve (AUC)
Nicotine pharmacokinetics with respect to initiation of in-clinic investigational product (IP) use following a 12-hour tobacco and nicotine abstinence | -5, -0.5, 3, 5, 7.5, 10, 15, 20, 30, 45, 60, 75, 90, 120, 150, 180, 240, 300, 360 minutes
  Determine maximum plasma nicotine concentration (Cmax), baseline adjusted
Nicotine pharmacokinetics with respect to initiation of in-clinic investigational product (IP) use following a 12-hour tobacco and nicotine abstinence | -5, -0.5, 3, 5, 7.5, 10, 15, 20, 30, 45, 60, 75, 90, 120, 150, 180, 240, 300, 360 minutes
  Determine maximum plasma nicotine concentration (Tmax)
Subjective effects scores for Urge to Smoke (UTS) | Three times during baseline UB cigarette smoking and 3 times per day for 5 days after switch to randomized IP use
  Determine trends in Urge to Smoke
Changes in biomarkers of tobacco exposure after a 5-day, in-clinic switch from usual brand (UB) cigarettes to an Electronic Cigarette or Nicotine Gum | 6 days
  Determine trends in plasma nicotine and cotinine during randomized IP use compared to UB smoking
Changes in biomarkers of tobacco exposure after a 5-day, in-clinic switch from usual brand (UB) cigarettes to an Electronic Cigarette or Nicotine Gum | 6 days
  Determine percent change in urinary total nicotine equivalents (Nicotine + 10 metabolites), after 5 days of randomized IP use compared to UB smoking
Changes in biomarkers of tobacco exposure after a 5-day, in-clinic switch from usual brand (UB) cigarettes to an Electronic Cigarette or Nicotine Gum | 6 days
  Determine percent change in urinary nitrosamines and metabolites, after 5 days of randomized IP use compared to UB smoking
Changes in biomarkers of tobacco exposure after a 5-day, in-clinic switch from usual brand (UB) cigarettes to an Electronic Cigarette or Nicotine Gum | 6 days
  Determine percent change in urinary 3-aminobiphenyl, after 5 days of randomized IP use compared to UB smoking
Changes in biomarkers of tobacco exposure after a 5-day, in-clinic switch from usual brand (UB) cigarettes to an Electronic Cigarette or Nicotine Gum | 6 days
  Determine percent change in urinary 4-aminobiphenyl, after 5 days of randomized IP use compared to UB smoking
Changes in biomarkers of tobacco exposure after a 5-day, in-clinic switch from usual brand (UB) cigarettes to an Electronic Cigarette or Nicotine Gum | 6 days
  Determine percent change in urinary 1-aminonaphthalene, after 5 days of randomized IP use compared to UB smoking
Changes in biomarkers of tobacco exposure after a 5-day, in-clinic switch from usual brand (UB) cigarettes to an Electronic Cigarette or Nicotine Gum | 6 days
  Determine percent change in urinary 2-aminonaphthalene, after 5 days of randomized IP use compared to UB smoking
Changes in biomarkers of tobacco exposure after a 5-day, in-clinic switch from usual brand (UB) cigarettes to an Electronic Cigarette or Nicotine Gum | 6 days
  Determine percent change in urinary o-toluidine, after 5 days of randomized IP use compared to UB smoking
Changes in biomarkers of tobacco exposure after a 5-day, in-clinic switch from usual brand (UB) cigarettes to an Electronic Cigarette or Nicotine Gum | 6 days
  Determine percent change in urinary S-phenyl mercapturic acid, after 5 days of randomized IP use compared to UB smoking
Changes in biomarkers of tobacco exposure after a 5-day, in-clinic switch from usual brand (UB) cigarettes to an Electronic Cigarette or Nicotine Gum | 6 days
  Determine percent change in urinary 1-hydroxypyrene, after 5 days of randomized IP use compared to UB smoking
Changes in biomarkers of tobacco exposure after a 5-day, in-clinic switch from usual brand (UB) cigarettes to an Electronic Cigarette or Nicotine Gum | 6 days
  Determine percent change in urinary 3-hydroxy-benzo[a]pyrene, after 5 days of randomized IP use compared to UB smoking
Changes in biomarkers of tobacco exposure after a 5-day, in-clinic switch from usual brand (UB) cigarettes to an Electronic Cigarette or Nicotine Gum | 6 days
  Determine percent change in urinary 1-hydroxynapthalene, after 5 days of randomized IP use compared to UB smoking
Changes in biomarkers of tobacco exposure after a 5-day, in-clinic switch from usual brand (UB) cigarettes to an Electronic Cigarette or Nicotine Gum | 6 days
  Determine percent change in urinary 2-hydroxynaphthalene, after 5 days of randomized IP use compared to UB smoking
Changes in biomarkers of tobacco exposure after a 5-day, in-clinic switch from usual brand (UB) cigarettes to an Electronic Cigarette or Nicotine Gum | 6 days
  Determine percent change in urinary 2-hydroxyfluorene, after 5 days of randomized IP use compared to UB smoking
Changes in biomarkers of tobacco exposure after a 5-day, in-clinic switch from usual brand (UB) cigarettes to an Electronic Cigarette or Nicotine Gum | 6 days
  Determine percent change in urinary N-acetyl-S-(3-amino-3-oxypropyl) cysteine, after 5 days of randomized IP use compared to UB smoking
Changes in biomarkers of tobacco exposure after a 5-day, in-clinic switch from usual brand (UB) cigarettes to an Electronic Cigarette or Nicotine Gum | 6 days
  Determine percent change in urinary N-acetyl-S-(3-amino-2-hydroxy-3-oxopropyl) cysteine, after 5 days of randomized IP use compared to UB smoking
Changes in biomarkers of tobacco exposure after a 5-day, in-clinic switch from usual brand (UB) cigarettes to an Electronic Cigarette or Nicotine Gum | 6 days
  Determine percent change in urinary 3-hydroxypropyl mercapturic acid, after 5 days of randomized IP use compared to UB smoking
Changes in biomarkers of tobacco exposure after a 5-day, in-clinic switch from usual brand (UB) cigarettes to an Electronic Cigarette or Nicotine Gum | 6 days
  Determine percent change in urinary 3-hydroxy-1-methylpropyl-mercapturic acid, after 5 days of randomized IP use compared to UB smoking
Changes in biomarkers of tobacco exposure after a 5-day, in-clinic switch from usual brand (UB) cigarettes to an Electronic Cigarette or Nicotine Gum | 6 days
  Determine percent change in urinary monohydroxybutyl mercapturic acid, after 5 days of randomized IP use compared to UB smoking
Changes in biomarkers of tobacco exposure after a 5-day, in-clinic switch from usual brand (UB) cigarettes to an Electronic Cigarette or Nicotine Gum | 6 days
  Determine percent change in urinary 2-cyanoethyl mercapturic acid, after 5 days of randomized IP use compared to UB smoking
Changes in biomarkers of tobacco exposure after a 5-day, in-clinic switch from usual brand (UB) cigarettes to an Electronic Cigarette or Nicotine Gum | 6 days
  Determine percent change in urinary 2-hydroxyethyl mercapturic acid, after 5 days of randomized IP use compared to UB smoking
Changes in biomarkers of tobacco exposure after a 5-day, in-clinic switch from usual brand (UB) cigarettes to an Electronic Cigarette or Nicotine Gum | 6 days
  Determine percent change in urinary thiocyanate, after 5 days of randomized IP use compared to UB smoking
Changes in biomarkers of tobacco exposure after a 5-day, in-clinic switch from usual brand (UB) cigarettes to an Electronic Cigarette or Nicotine Gum | 6 days
  Determine percent change in urinary mutagenicity, after 5 days of randomized IP use compared to UB smoking

SECONDARY OUTCOMES:
Daily product use amounts | Daily during baseline UB cigarette smoking and each day for 5 days after switch to randomized IP use

CONTACTS AND LOCATIONS:
Overall Officials: Harry Alcorn, Jr., PharmD, Principal Investigator — Davita Clinical Research
Locations (1):
- DaVita Clinical Research, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No